CLINICAL TRIAL: NCT03867994
Title: Comparison of Carvedilol and Atorvastatin for Prevention of Contrast-Induced Nephropathy After Cardiac Catheterization
Brief Title: Comparison of Carvedilol and Atorvastatin for Preventing of Contrast-Induced Nephropathy.
Acronym: CIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: rabab ahmed mohamed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, rabab ahmed mohamed, Teaching Assistant in clinical pharmacy department, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: beta-blockers and statins
Record Dates: First submitted 2019-01-14; First posted 2019-03-08 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Contrast-induced Nephropathy
Keywords: Cardiac catheterization, carvedilol, atorvastatin.
MeSH Terms: interventions — Atorvastatin; Carvedilol; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This prospective study is intended to evaluate if carvedilol has any potential protective effect over atorvastatin on the development of contrast-induced nephropathy (CIN) following cardiac catheterization in patients with moderate to high risk for CIN.
Who Masked: Participant
Masking Description: the patients were selected randomly and divided for three groups prospectively. the design was single-blinded randomized controlled study at which the researcher was aware by the allocation of the groups while the patients were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Experimental): included 49 patients who received high dose statin (80 mg atorvastatin) 12 hours before CC and 40 mg just before CC +hydration with saline (0.9% NaCl) at 0.5-1 mg/kg/hour for 4-6 hours before and 4-6 hours after cardiac catheterization.
  Interventions: Drug: Atorvastatin; Drug: saline
- Group (B) (Experimental): included 48 patients who received 12.5 mg carvedilol twice daily for 7 days before CC and continued for 24 hours after the CC +hydration with saline (0.9% NaCl) at 0.5-1 mg/kg/hour for 4-6 hours before and 4-6 hours after cardiac catheterization.
  Interventions: Drug: Carvedilol; Drug: saline
- Group (C) (Experimental): included 47 patients who did not receive any medications but only hydration with saline (0.9% NaCl) at 0.5-1 mg/kg/hour for 4-6 hours before and 4-6 hours after cardiac catheterization
  Interventions: Drug: saline

INTERVENTIONS:
Drug: Atorvastatin
  Arms: Group (A)
Drug: Carvedilol
  Arms: Group (B)
Drug: saline
  Other Names: 0.9%NaCl

SUMMARY:
This prospective study is intended to evaluate if carvedilol has any potential protective effect over atorvastatin on the development of contrast-induced nephropathy (CIN) following cardiac catheterization in patients with moderate to high risk for CIN.

DETAILED DESCRIPTION:
This study enrolled 150 patients planned for CC, and randomly assigned for one of the three groups. Group (A)include 49 patients who received two atorvastatin dose 80 mg 12 hours before CC and 40 mg just before CC. Group (B) include 48 patients who received 12.5 mg carvedilol twice daily for 7 days before CC and continue for 24hrs after the day of CC, Group (C) include 47 patients who only hydrated with saline. All included patients were hydrated with saline intravenous 0.9 sodium chloride (NaCl) at 0.5-1 mg/kg/hour for 4-6 hours before and 4-6 hours after cardiac catheterization. Serum creatinine(Scr), blood urea nitrogen (BUN) and estimated glomerular filtration rate were evaluated at the baseline and after 48 from CC. Serum neutrophil-associated lipocalin (NGAL) was evaluated after 4 hours from CC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 70 years.
* Serum creatinine ≤ 1.5 mg/dL.
* Using a moderate dose of atorvastatin (40 mg or equivalent dose of other statins).
* Moderate to high-risk for CIN.

Exclusion Criteria:

* Patients suffering from ST-segment elevation myocardial infarction (STEMI)
* Patients need for immediate cardiac catheterization
* Elevated liver enzymes (Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) three times the upper limit of normal).
* Active infection.
* Any contraindication to carvedilol, or atorvastatin.
* Patients on regular use of vitamins, minerals.
* Using medication with antioxidant properties e.g., beta-carotene, vitamin E, vitamin C, selenium, theophylline or N-acetyl cysteine 7 days prior to CC.
* Hemodynamically unstable patients (defined as abnormal or unstable blood pressure, especially hypotension (blood pressure less than 90/60 mm Hg).
* Patients who required dialysis.
* Pregnancy.
* Using of carvedilol in the past three months.
* Using a nephrotoxic agent in the past 48 hours or exposure to a contrast agent in the past 7 days prior to cardiac catheterization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
development of contrast induced nephropathy | 1. Serum creatinine baseline was measured from venous blood (before initiating the hydration) and 48 hours after the CC procedure.
  CIN :(defined as absolute rise in the baseline serum creatinine concentration by 0.5 mg/dL after 48 hours from CC).

SECONDARY OUTCOMES:
Estimated Glomerular filtration rate (eGFR) | on admission, and re-calculated 48 hours post CC using
  Cockcroft-Gault equation was used to calculate (eGFR)

OTHER OUTCOMES:
Blood urea nitrogen (BUN) | On admission, and re-calculated 48 hours post CC using
  BUN was assayed using modified Urease-Berthelot Method (Egyptian company of biotechnology, Cairo. Egypt)
Serum Neutrophil gelatinase - associated lipocalin (NGAL) Description: . NGAL was assayed by enzyme -linked immunosorbent assay ELISA (Glory Science Co., Ltd, CHINA). | Baseline was measured from venous blood before the initiation of hydration, and 4 hours after CC procedure.
  . NGAL was assayed by enzyme -linked immunosorbent assay ELISA (Glory Science Co., Ltd, CHINA).

IPD SHARING:
Plan to Share IPD: Yes
All medical history included medication and disease, in addition to our study outcomes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available from the time of publication